CLINICAL TRIAL: NCT00378651
Title: Differentiation Between Esophageal and Tracheal Intubation Utilizing Neck Auscultation
Brief Title: Use of the Stethoscope to Confirm Breathing Tube Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CETINA-2
Record Dates: First submitted 2006-09-19; First posted 2006-09-20 (Estimated); Last update posted 2007-12-19 (Estimated); Status verified 2007-12

CONDITIONS: Intubation, Endotracheal
Keywords: Intubation, Endotracheal; Anesthesia, General

INTERVENTIONS:
Procedure: Neck Auscultation

SUMMARY:
This study is intended to validate the use of neck auscultation with an electronic stethoscope during intubation to confirm tracheal tube placement.

It is hypothesized that the ability to confirm correct tube placement with this technique will be similar to that of the end-tidal CO2 monitor, the current gold-standard device for confirming tracheal intubation.

DETAILED DESCRIPTION:
Unrecognized esophageal intubation results in disastrous consequences. Fortunately, a variety of techniques have been cited to confirm placement of the endotracheal tube. However, even end-tidal CO2 monitoring, considered to be the gold standard, has been associated with false positive and false negative results. In addition, use of this monitor requires ventilation through the tube, resulting in gastric distention if the esophagus has been intubated.

When the lateral neck is auscultated during insertion of an endotracheal tube, there is a distinct difference between the sounds generated by a tube placed in the esophagus compared to a tube inserted into the trachea. Stethoscopes are readily available in any OR setting, and ventilation and release of cricoid pressure need not occur prior to confirmation of tube placement. However, this technique has yet to be validated.

A series of sounds heard at the lateral neck during both tracheal and esophageal intubation will be recorded using an electronic stethoscope. These sound files will be played to a group including both experienced and inexperienced intubators, who will be asked to identify which sounds represent tracheal and esophageal intubation. Overall accuracy will be determined for the group of listeners.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery requiring general anesthesia with endotracheal intubation

Exclusion Criteria:

* Anticipated difficult intubation
* Contraindication to esophageal intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23
Dates: Start 2006-09; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Group accuracy: Correct identification of tube placement based on series of 30 sound files

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Shuen Tan, BSc(Hon), MD, Principal Investigator — Department of Anesthesia, University of Manitoba; Chris Christodoulou, MBCHB, FRCPC, Principal Investigator — St. Boniface Hospital
Locations (1):
- St. Boniface General Hospital, Winnipeg, Manitoba, Canada